CLINICAL TRIAL: NCT01296997
Title: Influence of a Calcium Phosphate Supplementation on the Secretion of Incretins in Humans.
Brief Title: Calcium Phosphate and Incretins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Gerhard Jahreis, Prof. Dr. habil, University of Jena
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LSEP H45-10
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Healthy Men
Keywords: calcium phosphate; incretins; human study
MeSH Terms: interventions — calcium phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- calcium phosphate (Experimental)
  Interventions: Dietary Supplement: calcium phosphate
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: calcium phosphate — the subjects consumed for 3 weeks a bread enriched with 1 g pentacalcium phosphate per day
  Arms: calcium phosphate
Other: placebo — the subjects consumed a bread without pentacalcium phosphate
  Arms: placebo

SUMMARY:
The study was conducted to investigate the effect of a calcium phosphate supplementation on the secretion of incretins.

ELIGIBILITY:
Inclusion Criteria:

* healthy men

Exclusion Criteria:

* intake of dietary supplements and chronic diseases

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
secretion of incretins | 3 weeks

SECONDARY OUTCOMES:
concentration of minerals in plasma | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof. Dr., Principal Investigator — Friedrich-Schiller-University Jena, Institute of Nutrition, Department of Nutritional Physiology
Locations (1):
- Friedrich-Schiller-University Jena, Institute of Nutrition, Department of Nutritional Physiology, Jena, Thuringia, Germany

REFERENCES:
- [Derived] Trautvetter U, Kiehntopf M, Jahreis G. Postprandial effects of calcium phosphate supplementation on plasma concentration-double-blind, placebo-controlled cross-over human study. Nutr J. 2013 Mar 8;12:30. doi: 10.1186/1475-2891-12-30. PMID 23510513